CLINICAL TRIAL: NCT04176094
Title: Intensive Care Unit Resident Scheduling Trial
Acronym: InCURS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Christopher Parshuram, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 1744
Record Dates: First submitted 2019-10-04; First posted 2019-11-25 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Patient Safety; Well-being; Education
Keywords: health service and systems research; population health

STUDY DESIGN:
Intervention Model Description: A cluster-randomized crossover trial will compare 16h vs. 24h overnight schedules for residents completing an ICU rotation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 16 hour schedule (Experimental): All residents assigned to an ICU randomized to a 16h overnight schedule will complete 16h overnight calls not preceded by an 8h daytime shift.
  Interventions: Other: 16h overnight duty; Other: Handover training
- 24 hour schedule (Active Comparator): All residents assigned to an ICU randomized to a 24h overnight schedule will complete 24h shifts when scheduled for overnight calls (8h daytime shift followed by a 16h overnight call).
  Interventions: Other: 24h overnight duty; Other: Handover training

INTERVENTIONS:
Other: 16h overnight duty — schedule observed by participating ICUs.
  Arms: 16 hour schedule
Other: 24h overnight duty — schedule observed by participating ICUs.
  Arms: 24 hour schedule
Other: Handover training — Formal handover training for residents in both interventions. ICUs with a pre-existing standardized handover training and process will be asked to continue handover practices throughout the study. In ICUs without a pre-existing standardized handover training and process, ICU education directors will be provided with materials to include in orientation of residents to the ICU and local training to ICU staff physicians at least once per year.

SUMMARY:
Many patients, doctors and others worry that tired doctors provide worse patient care, may not learn well and become burnt-out. In response to these concerns, some countries changed their laws to limit work-hours for doctors in training ('residents').

In Canada, most residents work six or seven 24-30h shifts each month. A recent Canadian report ordered by Health Canada said that making good decisions about resident work-hour rules was "significantly limited by quality evidence, especially evidence directly attributable to the Canadian context." Creating this evidence is the main goal of this research.

The pilot study in 2 intensive care units(ICU) found that shorter shifts may be worse for patients, and for residents were more tiring than expected but improved wellbeing. Learning was not assessed. Previous studies on resident work-hours report similar findings: conflicting effects for patients, benefits for resident wellbeing, inconsistent and under-studied effects on learning. Overall, these results are not conclusive and confirm the need for a larger study.

The current study will provide high-quality Canadian evidence. The investigators will compare two common ICU schedules used in Canada: resident shifts of 16h and 24h. ICU patients are very sick, there is little margin for error: they need doctors who know them well and are thinking clearly.

The effects of each schedule on patients and residents will be measured. For patients, mortality rates and harm caused by care in ICU will be studied. For resident education, their learning about managing common illnesses in ICU, to do basic ICU procedures, and communicate with families will be studied. For resident wellbeing measures will include sleepiness, other fatigue symptoms, and burnout.

Investigators will study both resident and patient outcomes so that Canadians can understand trade-offs linked to changing schedules. With this knowledge, Canadians can expect safer care for today's patients and better-trained doctors for the patients of tomorrow.

DETAILED DESCRIPTION:
Background: Strategies to manage residents' fatigue must balance patient safety, resident education and resident wellbeing. The trade-offs among these are not fully understood. A Canadian cluster-randomized clinical trial will provide urgently needed evidence to inform resident scheduling practice and policy.

Previous work questions assumptions used to justify duty hour reduction. The investigators found residents working overnight are fatigued but do sleep, are not chronically sleep deprived, learn effectively immediately after being 'on-call' and learn in a 4-week ICU rotation. The pilot cluster randomized clinical trial of 12, 16 and 24h overnight duty suggests that patient safety is compromised with duty periods shorter than 24h: more harmful errors occurred in the 12h schedule, and residents' knowledge of patients and clinical decisions were worst in the 16h schedule. Mortality was similar. Resident wellbeing was worst in the 24h schedule, suggesting a trade-off between patient safety and resident wellbeing. Education was not assessed.

The 8 other randomized clinical trials of physician schedules are from the US; 2 studied residents (the providers of first line overnight medical care in Canadian hospitals), and 6 had low power for important effects on patient outcomes. None found differences in mortality or harmful errors or robustly examined educational outcomes.

With Canadian Institutes of Health Research bridge funding the investigators completed a Canada-wide survey showing that most ICU overnight in-house physician staffing is by residents, and a pilot of education outcomes demonstrating the feasibility, responsiveness and discriminative power of competency assessment.

Goals: To evaluate the effects of 16h and 24h resident duty schedules on patient mortality and safety, resident education and resident wellbeing.

Design: A cluster-randomized crossover trial will compare 16h vs. 24h overnight schedules for residents rotating to ICU. Eligible ICUs will care for adult patients, and are anticipated to have rotating residents performing overnight in-house duty.

Intervention: 16h and 24h overnight schedules will both be applied for 52 weeks at each site. Schedule crossover order will be randomly allocated (1:1 ratio). All in-house residents will participate in the schedule.

Consent will be obtained for resident measurements.

Outcomes: are in 3 domains, Patient, Resident Education and Resident Wellbeing. The primary outcome is hospital mortality to 90 days following index ICU admission. Mortality is objective, patient-relevant, frequent (12-20% in adult ICU) and reflects the quality and safety of care. The main resident education outcome is cognitive reasoning, and the main resident wellbeing outcome is emotional exhaustion.

Study of patients and residents in 18 ICUs has power >90% for a 2% difference in mortality and of 90% for important differences in resident education and resident wellbeing. Analyses will use hierarchical regression models to account for clustering by ICU.

Expertise: The research team includes experts in patient safety, postgraduate medical education, randomized clinical trials, sleep, and 2 national-level decision-makers.

Impact: Key stakeholders actively seek high-quality data about the effects of common overnight schedules on patients and residents. Understanding the benefits and trade-offs will support creation of evidence informed policy about resident schedules and mitigation strategies. This knowledge will improve care for patients and help better train doctors.

ELIGIBILITY:
Inclusion Criteria for ICUs:

* Admit adult patients (≥18 years);
* Are anticipated to have sufficient rotating residents from Royal College of Physicians and Surgeons of Canada -accredited training programs to provide overnight in-house coverage for at least 20 overnight periods in 28 days; and
* Are willing to participate in the study (schedule randomization, measurements).

Inclusion Criteria for Patients:

• Patients admitted to ICU during either period of the study.

Inclusion Criteria for Residents:

* Are enrolled in an accredited specialty training program of the Royal College of Physicians and Surgeons of Canada (internal or emergency medicine, surgery, anaesthesia, other, but not critical care medicine),
* Are able to perform overnight in-house duty with supervision from critical care trainees and intensivists, and
* Have the first 4 weeks of their ICU rotation entirely in one period. Residents who have participated in the study previously will not complete the competency assessments, however will be eligible to participate in the wellbeing and description of learning activities.

Inclusion Criteria for Supervisors:

• Are Physicians responsible for the supervision of residents and other trainees in the ICU, and include Critical Care Trainees and Staff Physicians.

Inclusion Criteria for ICU frontline staff:

• Are Registered nurses, registered respiratory therapists, pharmacists, social workers, physiotherapists and occupational therapists, who provide care in the ICU.

Exclusion Criteria for ICUs:

* ICUs with no rotating residents performing overnight in-house duty.
* ICUs that are anticipating a major change in ICU staffing (e.g. in-house intensivist added or removed, in-house fellow added or removed) or
* Are unwilling to have either resident schedule randomized, to provide study measurements or both.

Exclusion Criteria for Patients:

• Patients will be excluded if they are in the ICU at the start of a study period.

Exclusion Criteria for Residents:

* Residents enrolled in a critical care medicine accredited specialty training program,
* Who are not able to perform overnight in-house duty,
* Where the first 4 weeks of their ICU rotation are not in one period,
* Where the length of their ICU rotation is less than 4 week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Patient Mortality After Index ICU Admission (First ICU Admission within the study periods) | Up to 90 days following index ICU admission
  Rate of Hospital mortality to 90 days following index ICU admission. Patients discharged from hospital before 90 days will be assumed to be alive at 90 days.
Resident Cognitive Reasoning-Script Concordance Test | During 4th week of ICU rotation
  A Script Concordance Test will be administered in week 4 of the ICU resident rotation. Scoring was derived by administering the Script Concordance Test to an expert panel. The higher the overall rating for a resident, the closer their responses align with the expert panel. The minimum score is 0 and the maximum is 35.
Resident Burnout - Emotional Exhaustion | 4th week of ICU rotation
  The Emotional Exhaustion sub-scale of the Maslach Burnout Inventory will be measured in week four of the residents ICU rotation. Lower scores mean less emotional exhaustion, higher scores mean more emotional exhaustion. The lowest score is 0 and the highest score is 54.

SECONDARY OUTCOMES:
Rate of ICU Mortality | Measured daily from ICU admission to ICU discharge. Estimated average is 7 days.
  Patient death occurring during ICU admission.
Rate of Patient Adverse Events | During ICU stay and up to 3 days post ICU discharge
  Unplanned injury arising as a consequence of medical care during the time the patient was in the ICU that is associated with morbidity, requires treatment, prolongs hospital stay, or results in disability at discharge.
Rate of Medication Error | During ICU stay and up to 3 days post ICU discharge
  Reported or documented: dosing errors, wrong medication, or drug given to wrong patient.
Resident Procedural Competencies: Basic Airway Management | During 4th week of ICU rotation
  End-rotation simulation. Procedural skills will be assessed using the Objective Structured Assessment of Technical Skills Global Rating Scale. The scale measures 7 domains, including the participant's knowledge of instruments, respect for tissue, and knowledge of the procedure.
  Sub-scale ratings are averaged to create a global score: 1 is the minimum score and indicates the lowest performance; 5 is the maximum score and indicates the highest performance.
Resident Procedural Competencies: Central Venous Line | Week 4 of ICU rotation
  End-rotation simulation. Procedural skills will be assessed using the Objective Structured Assessment of Technical Skills Global Rating Scale. The scale measures 7 domains, including the participant's knowledge of instruments, respect for tissue, and knowledge of the procedure.
  Sub-scale ratings from 1 to 5 are averaged to create a global score: 1 is the minimum score and indicates the lowest performance; 5 is the maximum score and indicates the highest performance.
Resident Communication Competency | Week 4 of ICU rotation
  End-rotation simulation. Assessment of communication skills during a goals of care discussion with a simulated family member using a communication Analytic Global Rating Scale (AGRS). The scale will be used to assess 5 domains of the participant's communication: empathy, verbal expression, degree of coherence in the interview, non-verbal expression and an overall assessment of knowledge and skills.
  The sub-scale ratings are averaged to create a global score: 1 is the minimum score and indicates the lowest performance; 5 is the maximum score and indicates the highest performance.
Resident Depersonalization | Week 4 of ICU rotation
  The Maslach Burnout Inventory Depersonalization sub-scale will be used at week 4 of the resident ICU rotation. The range of scores is from 0 to 30. Higher scores indicate greater degrees of depersonalization. Lower scores indicate less depersonalization.
Resident Personal Accomplishment | Week 4 of ICU rotation
  The Maslach Burnout Inventory Personal Accomplishment sub-scale will be used at week 4 of the resident ICU rotation. The range of scores is from 0 to 48. Lower scores indicate less personal accomplishment. Higher scores indicate more personal accomplishment.
Resident Health Rating | Twice per week during the first 4 weeks of a residents ICU rotation
  Residents will rate their health on the day of survey. A score of 0 (the lowest value) represents the worst health and a score of 100 (the highest value) represents the best health the respondent can imagine.
Resident Nighttime Sleepiness | Two days per week at 8pm, midnight and 4am during the first 4 weeks of a residents ICU rotation
  Assessment of resident nighttime sleepiness using the Stanford Sleepiness Scale. The scale allows participants to indicate their level of sleepiness from on a 7-point scale from 1 to 7. A rating of 1 represents the least sleepy (most awake) and a rating of 7 the most sleepy. An additional (8th) response " I was asleep at the time of the assessment" is used if the resident was asleep at the time of the assessment.
Resident Daytime Sleepiness | Two days per week at 8am, noon and 4pm during the first 4 weeks of a residents ICU rotation
  Assessment of resident daytime sleepiness using the Stanford Sleepiness Scale. The scale allows participants to indicate their level of sleepiness from on a 7-point scale from 1 to 7. A rating of 1 represents the least sleepy (most awake) and a rating of 7 the most sleepy. An additional (8th) response " I was asleep at the time of the assessment" is used if the resident was asleep at the time of the assessment.

OTHER OUTCOMES:
Rate of Patient ICU Re-admission | 48 hours post-ICU discharge
  Patient ICU Re-admission within 48hrs of ICU discharge.
Rate of Patient Treated Cardiac Arrest | During ICU stay and up to 3 days post ICU discharge
  Documented cessation of circulation. Cardiac compressions and/or defibrillation provided in the ICU.
  The measurement tool used is a study specific case report form (CRF).
Rate of Patient Bleeding | During ICU stay and up to 3 days post ICU discharge
  Major new bleed with laboratory evidence and requiring transfusion. Clinically important minor new bleed (not requiring transfusion).
  The measurement tool used is a study specific case report form (CRF).
Rate of Patient Thrombosis/Embolism | During ICU stay and up to 3 days post ICU discharge
  New, documented thrombosis or embolism confirmed with imaging. The measurement tool used is a study specific case report form (CRF).
Rate of Patient Cutaneous Injury | During ICU stay and up to 3 days post ICU discharge
  Documented new cutaneous injury requiring start or modification of treatment. The measurement tool used is a study specific case report form (CRF).
Rate of Patient Acquired Neurologic Injury | During ICU stay and up to 3 days post ICU discharge
  Documented new neurologic injury (motor/sensory deficit) and brain/spine imaging showing ischemic/haemorrhagic injury or documented peripheral nerve injury diagnosed by nerve testing/clinical examination.
  The measurement tool used is a study specific case report form (CRF).
Rate of Patient Central Line or Endotracheal Tube Loss | During ICU stay and up to 3 days post ICU discharge
  Unplanned loss of central line, arterial line, endotracheal tube, chest tube or Extracorporeal Membrane Oxygenator therapy cannula.
  The measurement tool used is a study specific case report form (CRF).
Rate of Patient Adverse Drug Events | During ICU stay and up to 3 days post ICU discharge
  Documented or suspected drug-related event. Drug(s) administered during ICU admission.
  The measurement tool used is a study specific case report form (CRF).
Rate of Patient Acquired Infection | During ICU stay and up to 3 days post ICU discharge
  diagnosis of infection, documented infection (positive culture), antibiotics started/changed and continued for at least 3 days or until death.
  The measurement tool used is a study specific case report form (CRF).
ICU Resource Utilization: Length of Stay | Measured daily from the date of ICU admission to the date of ICU discharge for each enrolled patient. Estimated average is 7 days.
  Number of whole or part calendar days a patient spends in the ICU. The measurement tool used is a study specific case report form (CRF).
ICU Resource Utilization: Duration of Mechanical Ventilation | From the date of a patients ICU admission to the date of that patient's ICU discharge. Estimated average is 7 days.
  Number of whole or part calendar days of mechanical ventilation a patient received while in the ICU.
  The measurement tool used is a study specific case report form (CRF).
ICU Resource Utilization: Duration of Acute dialysis | From the date of a patients ICU admission to the date of that patient's ICU discharge. Estimated average is 7 days.
  Number of whole or part calendar days of acute dialysis a patient received while in the ICU.
  The measurement tool used is a study specific case report form (CRF).
ICU Resource Utilization: Duration of Inhaled Pulmonary Vasodilators | From the date of a patients ICU admission to the date of that patient's ICU discharge. Estimated average is 7 days.
  Number of whole or part calendar days of inhaled pulmonary vasodilators a patient received while in the ICU.
  The measurement tool used is a study specific case report form (CRF).
ICU Resource Utilization: Duration of Mechanical Circulatory Support | From the date of a patients ICU admission to the date of that patient's ICU discharge. Estimated average is 7 days.
  Number of whole or part calendar days of mechanical circulatory support a patient received while in the ICU.
  The measurement tool used is a study specific case report form (CRF).
ICU Resource Utilization: Duration of Inotrope-vasoactive therapy | From the date of a patients ICU admission to the date of that patient's ICU discharge. Estimated average is 7 days.
  Number of whole or part calendar days of inotrope-vasoactive therapy a patient received while in the ICU.
  The measurement tool used is a study specific case report form (CRF).
ICU Resource Utilization: Duration of non-invasive mechanical ventilation | From the date of a patients ICU admission to the date of that patient's ICU discharge. Estimated average is 7 days.
  Number of whole or part calendar days of non-invasive mechanical ventilation therapy a patient received while in the ICU.
  The measurement tool used is a study specific case report form (CRF).
Resident Daily Activities | Twice per week during the first 4 weeks of a residents ICU rotation
  Residents will be asked to indicate the learning activities they participated in while on duty.
  The measurement tool used is a study specific case report form (CRF).
Resident Wellbeing: Weekly Description | During the first 4 weeks of a residents ICU rotation
  Weekly questionnaire to describe the number of times residents were: exposed to bodily fluids, were the subject of inappropriate personal comments, received physical threats.
  The measurement tool used is a study specific case report form (CRF).
Resident Perception of Learning Climate | Week 4 of ICU rotation
  End-of-rotation survey using the Dutch Residency Educational Climate Test. The Dutch Residency Educational Climate Test is to describe the resident's opinion regarding: Educational atmosphere, teamwork, role of ICU attending physicians, coaching and assessments, resident peer collaboration, adaptability of work to resident's competence, accessibility of supervisors, formal education and patient site out. Each section will be rated from 1= strongly disagree to 5=strongly agree. The higher the score, the better the learning climate. The maximum score is 175 the minimum score is 35.
Duration of Resident sleep | During 7 days of the ICU rotation
  On-duty sleep, pre-duty sleep, post-duty sleep measured in hours and minutes by actigraphy
Rate of Resident Needle Stick Injuries | During 4 weeks of ICU
  Weekly questionnaire to describe the number of times residents experienced a needle-stick injury or other unintended bodily fluid exposure.
  The measurement tool used is a study specific case report form (CRF).
Resident Motor Vehicle Collisions | Each Week of ICU rotation. Average duration 4 weeks.
  Weekly questionnaire to capture the number of times residents were experienced crashes/near crashes.
  The measurement tool used is a study specific case report form (CRF).
Supervising Physician Workload | Twice per week for duration of the study for 2 years at each site.
  Survey of supervising staff perceived workload will be completed twice per week. Questions include the number of times the supervising staff communicated with the resident during overnight duty, their departure time from the ICU, and the number of times they returned to ICU overnight.
  The measurement tool used is a study specific case report form (CRF).
Supervising Physician Perceptions of resident performance | Twice per week for duration of the study for 2 years at each site.
  Survey of supervising staff perceived resident performance (quality of diagnosis, quality of management and occurrence of medical errors).
  The measurement tool used is a study specific case report form (CRF).
Amount of Sleep in last 12 hours. | Twice per week during the first 4 weeks of a residents ICU rotation
  Residents will be asked to report the number of hours the slept in the 12 hours before they started work. The minimum will be zero hours and the maximum will be 12 hours.
Number of Resident Symptoms in last 24 hours. | Twice per week during the first 4 weeks of a residents ICU rotation
  Residents will describe the presence of each of 14 physical symptoms they experienced in the 24 hours prior to measurement. The measurement tool used is a study specific case report form (CRF). The minimum is 0 symptoms, the maximum is 14 symptoms. A greater number of reported symptoms is worse. A smaller number of reported symptoms is better.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Parshuram, MD, Principal Investigator — The Hospital for Sick Children; Dominique Piquette, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (5):
- Canada (5):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parshuram CS, Amaral AC, Ferguson ND, Baker GR, Etchells EE, Flintoft V, Granton J, Lingard L, Kirpalani H, Mehta S, Moldofsky H, Scales DC, Stewart TE, Willan AR, Friedrich JO; Canadian Critical Care Trials Group. Patient safety, resident well-being and continuity of care with different resident duty schedules in the intensive care unit: a randomized trial. CMAJ. 2015 Mar 17;187(5):321-9. doi: 10.1503/cmaj.140752. Epub 2015 Feb 9. PMID 25667258